CLINICAL TRIAL: NCT01323010
Title: Efficacy and Safety of Increasing Doses of Inhaled Albuterol Administered by Metered Dose Inhalers in Children With Acute Wheezing Episodes
Brief Title: Efficacy and Safety of Increasing Doses of Inhaled Albuterol in Children With Acute Wheezing Episodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luiz Vicente Ribeiro Ferreira da Silva Filho, MD PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hidalba
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Asthma; Children
Keywords: asthma; albuterol; metered dose inhalers
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol - Experimental (Experimental): Albuterol dosages during the first hour include 900 mcg (up to 15 kg), 1200 mcg (> 15 to 20 kg), 1500 mcg (> 20 to 25 kg) and 1800 mcg (> 25 kg).
  Interventions: Drug: Albuterol - Experimental
- Albuterol - Control (Active Comparator): Albuterol dosages during the first hour include either 600 mcg (up to 25 kg) or 1200 mcg (> 25 kg).
  Interventions: Drug: Albuterol - Control

INTERVENTIONS:
Drug: Albuterol - Experimental — The Experimental group will receive higher doses of albuterol in the first hour: 900 mcg (up to 15 kg), 1200 mcg (> 15 to 20 kg), 1500 mcg (> 20 to 25 kg) and 1800 mcg (> 25 kg).
  Other Names: Ventolin
  Arms: Albuterol - Experimental
Drug: Albuterol - Control — The Control group will receive the following doses of albuterol in the first hour 600 mcg (up to 25 kg) or 1200 mcg (> 25 kg)
  Other Names: Ventolin
  Arms: Albuterol - Control

SUMMARY:
Metered dose inhalers with spacers are devices capable of providing higher rates of lung deposition of drugs such as beta agonists when compared to conventional nebulizers, but there is no consensus about the optimal dose when this is the device of choice and there is evidence that younger children need proportionally higher doses of albuterol (in μg/kg) when compared to older children. Other factors that may interfere with response to albuterol treatment include the genetics of the beta adrenergic receptor (ADRβ2) and infectious etiology of the wheezing attack. This study will assess the effectiveness of a dose regimen that prioritizes higher doses of albuterol, with doses in μg/kg higher for younger children. Security of this new dosing regimen will be assessed by monitoring clinical side effects and serum levels of albuterol, but the investigators will also examine the presence of 12 different respiratory viruses in these patients and evaluate the influence of ADRβ2 receptor genetics in the response to albuterol. The primary outcome measure will be the need for hospitalization. Secondary outcomes will include a change in clinical score, respiratory rate and forced expiratory volume in the first second, the need for additional treatments and length of stay in the emergency room for those not hospitalized.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blinded, controlled study. The patients will be randomly assigned to one of the treatment groups (experimental or control groups).

The patients will be assessed 1 hour later and every 30 minutes thereafter until discharge. Following 4 hours in the emergency room, any patient who do not meet the discharge criteria (PRAM score ≤ 3 and SpO2 ≥ 92%) will be admitted to the hospital. Each patient's attending physician will determine the need for additional therapies following the first hour.

Identification of respiratory viruses in the nasal lavage samples wil be performed using the CLART PneumoVir® kit.

Albuterol plasmatic levels will be analyzed via HPLC (High Performance Liquid Chromatography).

To genotype the ADBR2 receptor (blood samples), the gene regions encompassing the Arg16Gly, Gln27Glu, and Arg19Cys Thr164Ile polymorphisms will be amplified via PCR. The resultant amplimers were then sequenced.

A sample of 124 patients (62 in each group) was calculated to provide an 80% power with which to detect a significant difference of at least 30 minutes in the lengths of stay between the groups. The chi-square test will be used to compare hospital admission rates and tremor rates. For all other outcomes, t-tests for mean comparisons (variables with a normal distribution), a Mann Whitney test (nonparametric data) and ANOVA with repeated measures will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2 to 18 years;
2. History of two or more previous episodes of wheezing treated with bronchodilators in the last year;
3. Wheezing attacks characterized by coughing, difficulty breathing and auscultation of expiratory wheezing or prolonged expiration;
4. Intensity of wheezing attacks defined by PRAM score as moderate or severe (PRAM ≥ 5).

Exclusion Criteria:

1. Pre-existing chronic diseases such as bronchopulmonary dysplasia, cystic fibrosis, bronchiolitis obliterans or other chronic pulmonary or cardiovascular disease;
2. Initial clinical status indicating immediate ventilatory support, need for subcutaneous or intravenous bronchodilators;
3. Decreased level of consciousness;
4. Using a β-agonist in the four hours prior to arrival.
5. Use of corticosteroids in the last 24h.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Vicente RF Silva Filho, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto da Crianca HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Muchao FP, Souza AV, Souza JME, Silva Filho LVRFD. Association between beta-2 adrenergic receptor variants and clinical outcomes in children and adolescents with acute asthma. Einstein (Sao Paulo). 2022 Mar 25;20:eAO6412. doi: 10.31744/einstein_journal/2022AO6412. eCollection 2022. PMID 35352766
- [Derived] Muchao FP, Souza JM, Torres HC, De Lalibera IB, de Souza AV, Rodrigues JC, Schvartsman C, da Silva Filho LV. Albuterol via metered-dose inhaler in children: Lower doses are effective, and higher doses are safe. Pediatr Pulmonol. 2016 Nov;51(11):1122-1130. doi: 10.1002/ppul.23469. Epub 2016 May 12. PMID 27171324

RESULTS

PARTICIPANT FLOW:
Groups:
- Albuterol - Higher Dose (Experimental): Dosing will be individualized in four categories according to body weight
  Albuterol - Experimental: The Experimental group will receive higher doses of albuterol in the first hour: up to 15 kg of weight: 900 mcg; 15 to 20 kg: 1200 mcg; 20 to 25 kg: 1500; more than 25 kg: 1800 mcg
- Albuterol - Lower Dose (Control): Dosing will be dived according to consensus recommendations in only two categories according to body weight
  Albuterol - Control: The Control group will receive 600 mcg for those with weight under 25kg and 1200 mcg for those grater than 25 kg
Period: Overall Study
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Started | 60 | 59
Completed | 60 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: Dosing will be individualized in four categories according to body weight
  Albuterol - Experimental: The Experimental group will receive higher doses of albuterol in the first hour: up to 15 kg of weight: 900 mcg; 15 to 20 kg: 1200 mcg; 20 to 25 kg: 1500; more than 25 kg: 1800 mcg
- Control Group: Dosing will be dived according to consensus recommendations in only two categories according to body weight
  Albuterol - Control: The Control group will receive 600 mcg for those with weight under 25kg and 1200 mcg for those grater than 25 kg
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.68 (3.38) | 6.42 (3.74) | 6.55 (3.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 30 | 33 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 16 | 12 | 28
  More than one race | 32 | 34 | 66
  Unknown or Not Reported | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Hospital Admission
Description: Hospital admission was defined as the need to stay in the emergency room for more than 4 hours, due to the failure to meet the discharge criteria (PRAM score ≤ 3 and pulse oximetry, ≥ 92%)
Time Frame: Starting at 4 hours post-treatment
Measure: Number; unit: participants
Groups:
- Albuterol - Higher Dose (Experimental): Dosing was individualized in four categories according to body weight
  Albuterol - Experimental: The Experimental group received higher doses of albuterol in the first hour: up to 15 kg of weight: 900 mcg; 15 to 20 kg: 1200 mcg; 20 to 25 kg: 1500; more than 25 kg: 1800 mcg
- Albuterol - Lower Dose (Control): Dosing was dived according to consensus recommendations in only two categories according to body weight
  Albuterol - Control: The Control group received 600 mcg for those with weight under 25kg and 1200 mcg for those grater than 25 kg
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
participants | 11 | 8
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.689, Chi-squared

2. Secondary Outcome: Forced Expiratory Volume in the First Second
Description: Change in FEV1 one hour post-treatment in comparison with baseline. Spirometry was performed only in subjects older than 6 years and who could perform the maneuver properly.
Time Frame: One hour post-treatment in comparison with baseline
Measure: Mean (Standard Deviation); unit: percentage of predicted
Groups:
- Albuterol - Lower Dose (Control): Dosing was individualized according to consensus recommendations in only two categories according to body weight
  Albuterol - Control: The Control group received 600 mcg for those with weight under 25kg and 1200 mcg for those grater than 25 kg
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 18 | 12
percentage of predicted | 14.67 (16.62) | 11.3 (15.62)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.591, t-test, 2 sided

3. Secondary Outcome: Change in PRAM Score After One Hour
Description: Change in the Pediatric Respiratory Assessment Measure (PRAM) score one hour post-treatment in comparison with baseline.
  The PRAM score is used to assess the severity of asthma attacks, it ranges from 0 to 15, and the higher the score, the greater the severity of the attack.
  We calculated the difference between the PRAM score measured one hour post treatment and the PRAM score at baseline (PRAM score 1 hour - PRAM score baseline).
  The larger the absolute value of the difference, the better the outcome (e.g., a difference of -4 indicates a better outcome that a difference of -2).
  minimum value of the difference (Albuterol - Higher Dose, experimental group): -8 maximum value of the difference (Albuterol - Higher Dose, experimental group): 0
  minimum value of the difference (Albuterol - Lower Dose, control group): -8 maximum value of the difference (Albuterol - Lower Dose, control group): 0
Time Frame: One hour post-treatment
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
units on a scale | -3 [-5 to -2] | -4 [-5 to -3]
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.150, ANOVA; Method: ANOVA with repetead measures for non parametric data proposed by Brunner and Piri

4. Secondary Outcome: Albuterol Determination in the Plasma
Description: Albuterol determination in the plasma was carried out at at discharge or hospital admission (up to 4 hours post treatment), dosage was accomplished by High Performance Liquid Chromatography.
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment)
Population: It was possible to obtain albuterol plasma levels from 52 patients in the study group and 51 in the control group (in the other samples, this analysis was not feasible due to hemolysis).
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 52 | 51
ng/ml | 2.57 [0 to 15.8] | 1.08 [0 to 14.5]
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Changes in Glucose Serum Levels
Description: Changes in glucose serum levels at discharge or hospital admission (up to 4 hours post treatment) in comparison with baseline.
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment) in comparison with baseline.
Population: It was possible to obtain glucose serum levels from 57 patients in the study group and 55 in the control group (in the other samples, this analysis was not feasible due to hemolysis).
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 57 | 55
mg/dL | 34.73 (5.05) | 22.90 (5.25)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.108, ANOVA

6. Secondary Outcome: Electrocardiogram at Baseline
Description: Electrocardiogram performed at baseline
Time Frame: at baseline
Population: no electrocardiopraphic abnormalities were detected in both groups
Measure: Number; unit: participants with ECG abnormalities
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
participants with ECG abnormalities | 0 | 0

7. Secondary Outcome: Changes in Respiratory Rate After One Hour
Description: Change in respiratory rate one hour post-treatment in comparison with baseline.
Time Frame: One hour post-treatment in comparison with baseline
Measure: Mean (Standard Error); unit: breaths per minute
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
breaths per minute | -2.08 (1.03) | -4.31 (0.99)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.122, ANOVA

8. Secondary Outcome: Need for Additional Therapies
Description: The need for additional therapies such as magnesium sulphate or intravenous albuterol were recorded
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment)
Population: no patients received magnesium sulphate or intravenous albuterol in both groups
Measure: Number; unit: participants
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
participants | 0 | 0

9. Secondary Outcome: Changes in PRAM Score at Discharge or Hospital Admission
Description: Change in the Pediatric Respiratory Assessment Measure (PRAM) score at discharge or hospital admission (up to 4 hours post treatment) in comparison with baseline.
  The PRAM score is used to assess the severity of asthma attacks, it ranges from 0 to 15, and the higher the score, the greater the severity of the attack.
  We calculated the difference between the PRAM score measured at discharge or admission and the PRAM score at baseline (PRAM score discharge or admission - PRAM score baseline).
  The larger the absolute value of the difference, the better the outcome (e.g., a difference of -4 indicates a better outcome that a difference of -2).
  minimum value of the difference (Albuterol - Higher Dose, experimental group): -9 maximum value of the difference (Albuterol - Higher Dose, experimental group): 0
  minimum value of the difference (Albuterol - Lower Dose, control group): -9 maximum value of the difference (Albuterol - Lower Dose, control group): 1
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
units on a scale | -4.5 [-6 to -3] | -5 [-6 to -4]
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.164, ANOVA; Method: ANOVA with repetead measures for non paramteric data proposed by Brunner and Piri

10. Secondary Outcome: Changes in Potassium Serum Levels
Description: Changes in potassium serum levels at discharge or hospital admission (up to 4 hours post treatment) in comparison with baseline.
Time Frame: as for outcome 5
Population: It was possible to obtain potassium serum levels from 54 patients in the study group and 56 in the control group (in the other samples, this analysis was not feasible due to hemolysis).
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 54 | 56
mEq/L | -0.38 (0.10) | -0.59 (0.10)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.165, ANOVA

11. Secondary Outcome: Changes in Bicarbonate Serum Levels
Description: Changes in bicarbonate serum levels at discharge or hospital admission (up to 4 hours post treatment) in comparison with baseline.
Time Frame: as for outcome 5
Population: It was possible to obtain bicarbonate serum levels from 42 patients in the study group and 37 in the control group (in the other samples, this analysis was not feasible due to the long time to transport the samples to the laboratory in one of our centers).
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 42 | 37
mmol/L | -1.75 (0.26) | -1.44 (0.29)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.436, ANOVA

12. Secondary Outcome: Changes in Respiratory Rate at at Discharge or Hospital Admission.
Description: Changes in respiratory rate at discharge or hospital admission (up to 4 hours post treatment) in comparison with baseline.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: breaths per minute
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
breaths per minute | -2.92 (1.03) | -5.76 (0.99)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.046, ANOVA

13. Secondary Outcome: Change in Pulse Oximetry One Hour Post-treatment
Description: Change in pulse oximetry one hour post-treatment in comparison with baseline
Time Frame: One hour post-treatment in comparison with baseline
Measure: Mean (Standard Error); unit: percentage of oxygen saturation
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
percentage of oxygen saturation | 1.54 (0.29) | 1.39 (0.30)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.723, ANOVA

14. Secondary Outcome: Changes in Pulse Oximetry at Discharge or Hospital Admission.
Description: Changes in pulse oximetry at discharge or hospital admission (up to 4 hours post treatment) in comparison with baseline.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
percentage of oxygen saturation | 2.14 (0.32) | 1.59 (0.33)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.235, ANOVA

15. Secondary Outcome: Changes in Heart Rate After One Hour
Description: Change in heart rate one hour post-treatment in comparison with baseline.
Time Frame: One hour post-treatment in comparison with baseline
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
beats per minute | 1.75 (2.12) | -1.47 (2.12)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.284, ANOVA

16. Secondary Outcome: Changes in Heart Rate at Discharge or Hospital Admission
Description: Changes in heart rate at discharge or hospital admission (up to 4 hours post treatment) in comparison with baseline.
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment)
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
beats per minute | -0.263 (2.17) | -0.65 (2.17)
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.905, ANOVA

17. Secondary Outcome: Electrocardiogram One Hour Post-treatment.
Description: Electrocardiogram one hour post-treatment to identify possible rhythm disturbances.
Time Frame: One hour post-treatment
Population: No electrocardiographic abnormalities were detected im both groups
Measure: Number; unit: participants with ECG abnormalities
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
participants with ECG abnormalities | 0 | 0

18. Secondary Outcome: Electrocardiogram at Discharge or Hospital Admission
Description: Electrocardiogram at discharge or hospital admission to identify possible rhythm disturbances.
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment)
Population: No electrocardiographic abnormalities were detected in both groups.
Measure: Number; unit: participants with ECG abnormalities
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 60 | 59
participants with ECG abnormalities | 0 | 0

19. Secondary Outcome: Lengths of Stay in the Emergency Room
Description: lengths of stay in the emergency room for discharged patients
Time Frame: one to four hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Albuterol - Higher Dose (Experimental) | Albuterol - Lower Dose (Control)
Number analyzed (Participants) | 60 | 59
hours | 1.50 [1 to 2] | 1.40 [1 to 1.50]
Statistical Analysis 1: Comparison: Albuterol - Higher Dose (Experimental) vs Albuterol - Lower Dose (Control); Test type: Superiority or Other; p = 0.892, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Admission Rates in Patients With and Without Any Virus Detected
Description: Admission rates in patients with and without any of the following viruses detected by PCR in nasal lavage samples: Adenovirus; Bocavirus; Coronavirus; Enterovirus (Echovirus); Influenza (A H3N2, A H1N1/2009, B and C); Metapneumovirus (subtypes A and B); Parainfluenza 1, 2, 3 and 4 (subtypes A and B); Rhinovirus; Respiratory Syncytial Virus type A and Respiratory Syncytial Virus type B.
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment)
Population: We obtained nasal lavage samples from 117 individuals, in two patients it was not possible to collect nasal lavage samples.
Measure: Number; unit: percentage of participants
Groups:
- Virus Detected: patients with any virus detected by PCR
- No Virus Detected: patients with no virus detected by PCR
Arm/Group | Virus Detected | No Virus Detected
Number analyzed (Participants) | 73 | 44
percentage of participants | 12.3 | 22.7
Statistical Analysis 1: Comparison: Virus Detected vs No Virus Detected; Test type: Superiority or Other; p = 0.195, Chi-squared

21. Secondary Outcome: Admission Rates in Patients With and Without Rhinovirus Detect
Description: Admission rates in patients with and without rhinovirus detected by PCR in nasal lavage samples.
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment)
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Groups:
- Rhinovirus Detected: patients with rhinovirus detected by PCR
- No Rhinovirus Detected: patients with no rhinovirus detected by PCR
Arm/Group | Rhinovirus Detected | No Rhinovirus Detected
Number analyzed (Participants) | 49 | 68
percentage of participants | 10.2 | 20.6
Statistical Analysis 1: Comparison: Rhinovirus Detected vs No Rhinovirus Detected; Test type: Superiority or Other; p = 0.203, Chi-squared, Corrected

22. Secondary Outcome: Admission Rates in Patients With the Arg16Gly Polymorphisms
Description: Admission rates in patients with the Arg16Gly polymorphisms of the beta-2 adrenergic receptor (Arg16Gly, Arg16Arg and Gly16Gly genotypes).
Time Frame: at discharge or admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment)
Population: The sequencing of the beta-2 adrenergic receptor gene was performed in a subset of 60 patients, in the other samples these analysis were not feasible due to hemolysis.
Measure: Number; unit: participants
Groups:
- Arg16Gly Patients: Patients carrying the Arg16Gly genotype
- Gly16Gly Patients: Patients carrying the Gly16Gly genotype
- Arg16Arg Patients: Patients carrying the Arg16Arg genotype
Arm/Group | Arg16Gly Patients | Gly16Gly Patients | Arg16Arg Patients
Number analyzed (Participants) | 16 | 21 | 23
participants | 1 | 1 | 7
Statistical Analysis 1: Comparison: Arg16Gly Patients vs Gly16Gly Patients vs Arg16Arg Patients; Test type: Superiority or Other; p = 0.03, Chi-squared

ADVERSE EVENTS:
Time Frame: At discharge or hospital admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post-baseline).
Description: At discharge or hospital admission (up to 4 hours post-baseline, minimum 1 hour, maximum 4 hours) all possible adverse effects were monitored: significant changes in potassium and glucose and bicarbonate serum levels, electrocardiographic abnormalities or any clinical adverse effect.
  The last adverse event was detected 4 hours post-treatment.
Groups:
- Experimental Group: Dosing was individualized in four categories according to body weight
  Albuterol - Experimental: The Experimental group received higher doses of albuterol in the first hour: up to 15 kg of weight: 900 mcg; 15 to 20 kg: 1200 mcg; 20 to 25 kg: 1500; more than 25 kg: 1800 mcg
- Control Group: Dosing was dived according to consensus recommendations in only two categories according to body weight
  Albuterol - Control: The Control group received 600 mcg for those with weight under 25kg and 1200 mcg for those grater than 25 kg
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 36/60 | 37/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=60) | Control Group (N=59)
non symptomatic mild hypokalemia at discharge or hospital admission (up to 4 hours post-baseline). (Blood and lymphatic system disorders) | 7 (7) | 10 (10) — Non symptomatic mild hypokalemia in 17 patients, 10 in the control group, 7 in the experimental group. Only 2 patients showed values below 3.1 mEq/L. One patient in the experimental group: 2.8 mEq/L. One patient in the control group: 2.9mEq/L
non symptomatic mild hyperglycemia at discharge or hospital admission (up to 4 hours post-baseline) (Blood and lymphatic system disorders) | 29 (29) | 27 (27) — Non symptomatic mild hyperglycemia at discharge or hospital admission (up to 4 hours post treatment, minimum 1 hour, maximum 4 hours post treatment). No patients needed medical intervention.

LIMITATIONS AND CAVEATS:
The inclusion of a larger number of patients in this study may have uncovered differences in the efficacy outcomes studied between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No